CLINICAL TRIAL: NCT00999648
Title: Efficacy of Myofascial Trigger Point Pressure Release on Tinnitus Patients With Both Tinnitus and Myofascial Pain: a Double-blind Placebo Controlled Randomized Clinical Trial.
Brief Title: Efficacy of Myofascial Trigger Point Pressure Release on Tinnitus Patients
Acronym: MTP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Tinnitus Research Initiative (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Tanit Ganz Sanchez< MD, PhD, Departament of Otorhinolaryngology -University of Sao Paulo Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAPPesq 138306; TRI Grant /0704
Record Dates: First submitted 2009-10-21; First posted 2009-10-22 (Estimated); Last update posted 2009-10-22 (Estimated); Status verified 2009-10

CONDITIONS: Tinnitus; Myofascial Trigger Points
Keywords: Tinnitus; Myofascial Trigger Points; Myofascial Pain Syndrome; Controlled Clinical Trial
MeSH Terms: conditions — Tinnitus; Myofascial Pain Syndromes | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual therapy (Experimental): Myofascial trigger point pressure release
  Interventions: Other: Myofascial trigger point pressure release (deactivation)
- Control (Placebo Comparator): Placebo myofascial trigger point pressure release
  Interventions: Other: Placebo myofascial trigger point pressure release

INTERVENTIONS:
Other: Myofascial trigger point pressure release (deactivation) — The deactivation of MTP will be performed always by the same physiotherapist researcher using the same technique. Afterwards, a myofascial maneuver is performed in each treated muscle. All patients of the experimental group will be advised to perform complimentary procedures at home during the 10-week period treatment in order to maintain the status of the muscle up to the next session and to avoid losing the obtained result:(1) Stretching of the treated muscles, once a day for 25 seconds each, (2)Superficial heat in each treated muscle, once a day for 20 minutes, (3) Watch the correct postures during daily activities and sleeping.
  Other Names: Manual therapy, pressure release, digital pressure of MTP.
  Arms: Manual therapy
Other: Placebo myofascial trigger point pressure release — The physiotherapist researcher will press in an adjacent nontender muscle fibers of the same muscle that have MTP about 3cm to the right or to the left of each diagnosed MTP, using just a slight pressure on it, not enough for deactivation.
  Other Names: Placebo manual therapy
  Arms: Control

SUMMARY:
The objective of this study is to evaluate the efficacy of myofascial trigger (MTP) point deactivation for tinnitus control in a population with tinnitus and myofascial pain.

DETAILED DESCRIPTION:
A double blind placebo control randomized clinical trial was made to verify the efficacy of the treatment by deactivation of MTP, after 10 sessions, in tinnitus patients by means of comparison with a placebo treatment in a control group. Patients with tinnitus and frequent regional pain for at least 3 months in the head, neck and shoulder girdle were investigated in the Tinnitus Research Group of University of São Paulo Medical School. All of them underwent an interview with the otolaryngologist ("physician researcher"), an audiologist evaluation ("blind researcher"), another blind researcher evaluation for tinnitus and pain and a physiotherapist evaluation and randomization. Both blind researchers evaluated tinnitus and pain in the first, fifth and tenth session. The real treatment was made by a gradual and persistent digital pressure in each MTP previously diagnosed by the blind researcher (8 possible muscles) and some home orientations that included stretch, superficial heat in each treated muscle and watch the correct postures during daily activities and sleeping. In the control group physiotherapist researcher pressed in an adjacent non-tender muscle fibers of the same muscle that have MTP. No other complementary orientation was done.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects of any gender, age and race with presence of uni or bilateral tinnitus for at least 3 months;
2. Presence of pain complaint for at least 3 months in head, neck and shoulder girdle areas
3. Presence of at least one myofascial trigger point (MTP) related with the patient's pain complaint (active MTP).

Exclusion Criteria:

1. Pain complaint involving three or more quadrants of the body, regardless of its cause
2. Infiltration and/or specific treatment for deactivation of MTP in the last 6 months;
3. Use of medications or other techniques to treat tinnitus, pain or muscle disorders during the previous last month;
4. Impossibility of understanding the orientation and/or giving information during MTP evaluation (neurological or psychiatric diseases, bilateral severe or profound hearing loss, etc);
5. Absence of tinnitus perception during evaluation;
6. Pulsatile tinnitus or myoclonus (middle ear muscles or palatal myoclonus).
7. Tinnitus due to certain etiologies that require other specific types of treatment, determined according to the medical evaluation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory, tinnitus visual analogue scale (0 to 10), changes of numbers of sounds and frequency | first, fifth and tenth session of treatment

SECONDARY OUTCOMES:
Intensity and frequency of pain; number of active trigger point | first, fifth and tenth session of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Carina B. Rocha, PT, MA, Principal Investigator — University of Sao Paulo General Hospital
Locations (1):
- Clinics Hospital of University of Sao Paulo Medical School - Department of Otorhinolaryngology, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Rocha CA, Sanchez TG. Myofascial trigger points: another way of modulating tinnitus. Prog Brain Res. 2007;166:209-14. doi: 10.1016/S0079-6123(07)66018-X. PMID 17956784
- [Background] Bezerra Rocha CA, Sanchez TG, Tesseroli de Siqueira JT. Myofascial trigger point:a possible way of modulating tinnitus. Audiol Neurootol. 2008;13(3):153-60. doi: 10.1159/000112423. Epub 2007 Dec 13. PMID 18075244
- See also: Related Info — http://www.zumbido.org.br